CLINICAL TRIAL: NCT03330964
Title: Parallel Control Study of Electroacupuncture Stimulation the Acupoints of Yangming Channel on Prevention and Treatment of Oxaliplatin Neurotoxicity During the Peri-chemotherapy Period
Brief Title: Clinical Trial of Electroacupuncture Stimulation on Prevention and Treatment of Oxaliplatin Neurotoxicity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YJ-KY-2017-102
Record Dates: First submitted 2017-09-27; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-09

CONDITIONS: Neurotoxicity; Gastrointestinal Neoplasms
MeSH Terms: conditions — Neurotoxicity Syndromes; Gastrointestinal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electroacupuncture group (Experimental): The experimental group adopted chemotherapy combined with electro-acupuncture stimulated related acupoints for 3 days running.
  Interventions: Other: electro-acupuncture
- control group (No Intervention): The control group received chemotherapy only(same as the experimental group),but no electroacupuncture treatment.

INTERVENTIONS:
Other: electro-acupuncture — Electroacupuncture was administrated immediately after completion of oxaliplatin infusion,once a day for 3 days,30 minutes each time.
  Arms: electroacupuncture group

SUMMARY:
The clinical trail of electroacupuncture combined with oxaliplatin regimen on gastrointestinal carcinoma.This trail is randomized controled.Patients are diagnosed gastrointestinal cancer based on pathology or cell biology.They are randomized into 2 groups:both groups receive Oxaliplatin regimen.The treatment group receives electroacupuncture in addition to the chemotherapy.The control group only receive the same chemotherapy with the treatment group.Both group have the same adjuvant therapy.

DETAILED DESCRIPTION:
The clinical trail of electroacupuncture combined with oxaliplatin regimen on gastrointestinal carcinoma.This trail is randomized controled.Patients are diagnosed gastrointestinal cancer based on pathology or cell biology.They are randomized into 2 groups:both groups receive Oxaliplatin regimen.The treatment group receives electroacupuncture in addition to the chemotherapy.The control group only receive the same chemotherapy with the treatment group.Both group have the same adjuvant therapy.Mainly to study about oxaliplatin into electroacupuncture leads to the influence of the peripheral nerve toxicity.Other clinical evaluation includes chemotherapy drug toxicities,quality of life(QOL), etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80 ;
2. male and female ;
3. signed the informed consent form;
4. Eastern Cooperative oncology Group(ECOG)O-2,life expectancy more than 3 months;
5. Indication for Chemotherapy,no contraindication;
6. First time chemotherapy or at least 6 months after last chemotherapy and radiotherapy;
7. At least 8 weeks after last biotherapy;
8. Surgery:had not received transplantation surgery,at least 2 weeks after last major surgery.

Exclusion Criteria:

1. Chemotherapy is contraindicated;
2. Having the primary disease can cause the neuropathy;
3. A history of other malignant tumor in recent 5 years;
4. Less than 6 months after last chemotherapy or radiotherapy;
5. Less than 8 weeks after last biotherapy;
6. Being afraid of acupuncture seriously;
7. Had received transplantation surgery,less than 2 weeks after last major surgery;
8. Other researchers think is not suitable for this clinical trail.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Levi sensory nerve toxicity classification standard | every cycle of chemotherapy (measure 3 cycles, each cycle is 21 days), up to 3 months]
  Scoring scale

SECONDARY OUTCOMES:
The quality of life questionnaire(QLQ)-C30 | every cycle of chemotherapy (measure 3 cycles, each cycle is 21 days), up to 3 months]
  Scoring scale

OTHER OUTCOMES:
National Cancer Institute(NCI)Common Toxicity Criteria | every cycle of chemotherapy (measure 3 cycles, each cycle is 21 days), up to 3 months]
  Blood and Scoring scale

CONTACTS AND LOCATIONS:
Overall Officials: Xiaonan Cui, MD,PhD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University
Locations (2):
- China (2):
  - Oncology Department，The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning

IPD SHARING:
Plan to Share IPD: Undecided
Undecided